CLINICAL TRIAL: NCT03209778
Title: Involuntary Memories Investigation in Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The research was stopped because of recruitment difficulties at the end of the study due to a high drop-out rate for one of the two tasks included in the protocol.
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 6620
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Control participants without psychiatric nor neurological history
  Interventions: Other: Patients with Schizophrenia
- Patients with Schizophrenia (Experimental): Patients with schizophrenia or schizoaffective disorder according to DSM-V criteria
  Interventions: Other: Patients with Schizophrenia

INTERVENTIONS:
Other: Patients with Schizophrenia — Patients with schizophrenia or schizoaffective disorder according to DSM-V criteria

SUMMARY:
Patients with schizophrenia suffer from autobiographical memory disorders. Patients have difficulty to remember vividly personal past events when they are specifically asked for. Indeed, this task requires a good executive functioning to retrieve precise information stored in long term memory. Interestingly, executive functioning has been showed impaired in schizophrenia and studies showed that their autobiographical memory impairments were directed related to their executive dysfunction.

Yet, in daily life people remember more often autobiographical memories spontaneously, without trying voluntarily to recall them.

In that case, the involuntary recall of personal past events is much less sustained by executive functioning.

In this protocol the investigators would like to investigate and compare subjective characteristics of involuntary and voluntary autobiographical memories in order to highlight the role of executive dysfunction in patients' autobiographical memory impairments.

ELIGIBILITY:
Inclusion Criteria:

* - for patients only
* male or female
* age limits : 18-55 years old
* under the protection of health insurance
* who have signed up the consent form
* schizophrenia or schizo-affective disorder according to the DSM-5 criteria (APA, 2013).
* clinically stable for at least 2 months
* patients under guardianship or curatorship need agreement of their legal representative
* informed of the results of prior medical examination for controls only
* male or female
* age limits : 18-55 years old
* under the protection of health insurance
* who have sign up the consent form
* recruited from the general population and matched on gender, age years of schooling
* no psychiatric history (DSM-5)

Exclusion Criteria:

* for both patients and controls
* current severe or unstable somatic illness
* neurological history (brain injury > 15 minutes loss of consciousness , epilepsia, brain surgery…)
* current substance use disorder (DSM-5)
* current major depressive disorder (CDSS,BDI, HDRS)
* mental retardation (IQ < 70, WAIS-4, f-NART)
* history of general anesthesia 3 months prior to the experiment
* pregnancy declared by the subject
* breast feeding
* current legal control
* in emergency situation
* included during exclusion period in another experiment
* for controls only
* taking of antipsychotic drugs for the 3 weeks prior to inclusion
* under guardianship or curatorship

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Autobiographical subjective score taking into account memories vividness and specifity | 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No